CLINICAL TRIAL: NCT02465307
Title: Motion Analysis of Delirium in Intensive Care Units (ICUs) Subtitle 1: "ADAPT: Autonomous Delirium Monitoring and Adaptive Prevention"
Brief Title: Intelligent Intensive Care Unit
Acronym: ICU_Delirium
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400546 -N; 1750192 (Other Grant/Funding Number: National Science Foundation); 1R21EB027344-01 (NIH); R01NS120924-01 (NIH)
Record Dates: First submitted 2015-05-29; First posted 2015-06-08 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Delirium; Confusion
Keywords: Consciousness; Alertness; Cognition; Activity level; Delirium; Hyperactive delirium; Hypoactive delirium; Facial expression; Posture; Intensive care unit
MeSH Terms: conditions — Delirium; Confusion; Facial Expression | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Delirium group: ICU patients with a positive Confusion Assessment Method (CAM) score; observational using accelerometers, commercially available camera, and Internet Pod (iPod).
  Interventions: Behavioral: Confusion Assessment Method; Device: Accelerometer; Device: Commercially available camera; Device: Internet Pod (iPod)
- Control group: ICU patients with a negative Confusion Assessment Method (CAM) score; observational using accelerometers, commercially available camera, and Internet Pod (iPod).
  Interventions: Behavioral: Confusion Assessment Method; Device: Accelerometer; Device: Commercially available camera; Device: Internet Pod (iPod)
- Healthy control group: Healthy subjects that sleep in their home environment; observational using accelerometers, cortisol swabs, and Internet Pod (iPod)
  Interventions: Device: Accelerometer; Device: Internet Pod (iPod); Diagnostic Test: Cortisol Swab

INTERVENTIONS:
Behavioral: Confusion Assessment Method — Confusion Assessment Method (CAM) score
  Groups: Control group; Delirium group
Device: Accelerometer — 3 accelerometers (placed on upper arm, wrist and ankle) and 1 placed on wall as ambient light sensor
Device: Commercially available camera — As part of facial recognition video system
  Other Names: imaging
  Groups: Control group; Delirium group
Device: Internet Pod (iPod) — Monitors noise levels in the room
  Other Names: Sound detection
Diagnostic Test: Cortisol Swab — Cortisol level collected through self administered salivary swab
  Groups: Healthy control group

SUMMARY:
Delirium, as a common complication of hospitalization, poses significant health problems in hospitalized patients. Though about a third of delirium cases can benefit from intervention, detecting and predicting delirium is still very limited in practice. A common characterization of delirium is change in activity level, causing patients to become hyperactive or hypoactive which is manifested in facial expressions and total body movements. This pilot study is designed to test the feasibility of a delirium detection system using movement data obtained from 3-axis wearable accelerometers and commercially available camera with facial recognition video system in conjunction with electronics medical record (EMR) data to analyze the relation of whole-body movement and facial expressions with delirium.

DETAILED DESCRIPTION:
The aim of the study is to assess the potential of using motion and facial expression data to detect delirium in ICU patients by comparing motion and facial expression patterns in delirium and control groups. In this study, the investigators will use ActiGraph accelerometers to record each subject's movement patterns. Also, a processed video using a commercially available camera interfaces with a specialized program to identify patient facial expressions and movement patterns. A total of 60 participants will be enrolled with delirium, and 30 patients without delirium will be used as control group. Motion profiles will be compared in the motorically defined subgroups (hyperactive, hypoactive, normal) based on accelerometer and facial recognition data. Then, differences in facial expression, number of changes in postures, and percentage of time spent moving will be compared between motorically defined subgroups and in delirium and control groups. EMR data will also be used to assess the feasibility of detecting delirium by including additional information on related risk factors.

ELIGIBILITY:
Inclusion Criteria (ICU Patients):

* Intensive care unit patient
* 18 years of age or older

Exclusion Criteria (ICU Patients):

* Anticipated intensive care unit stay less than one day
* Less than 18 years of age
* Inability to wear a motion sensor watch (ActiGraph)

Inclusion Criteria (Healthy Controls):

* 18 years of age or older.
* sleeps in home environment

Exclusion Criteria (Healthy Controls):

* does not sleep in home environment
* Less than 18 years of age
* Inability to wear a motion sensor watch (ActiGraph)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU Patients: Patients who been hospitalized in an intensive care unit and have risk factors to develop delirium or delirium has been suspected by their medical provider.
  Healthy Controls: People who are healthy and sleep in their home environment.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
CAM/CAM-ICU | Changes from Baseline up to 7 Days
  Confusion Assessment Method for detection of delirium
Memorial Delirium Assessment Scale (MDAS) will be used for changes from baseline up to 7 days between the groups. | Changes from Baseline up to 7 Days
  MDAS denotes motor profile and defines motor subtyping. It has 10 items which assesses several areas of cognitive functioning (memory, attention, orientation and disturbances in thinking) and psychomotor activity. The items are rated on a four point scale (0-3) based on the current interaction with the patient or by assessment of behavior. A score of 13 shows the diagnosis of delirium.
Delirium Motor Subtyping Scale (DMSS-4) will be used for changes from baseline up to 7 days between the groups. | Changes from Baseline up to 7 Days
  Scoring from DMSS-4 which has 5 hyperactive and 8 hypoactive symptoms requires at least two symptoms to be present from either the hyperactive or hypoactive list to meet subtype criteria. The higher the score the higher the delirium.
Freedman Sleep Scale | Changes from Baseline up to 7 Days
  To determine sleep quality of patient for given day.

SECONDARY OUTCOMES:
Number of subjects who died | Baseline up to 7 Days
  Death at any time during admission
Number of subjects on mechanical ventilation | greater than 48 hours
  Number of subjects requiring mechanical ventilation greater than 48 hours.

OTHER OUTCOMES:
Facial amimia versus non-amimia expressions between the groups | Changes from Baseline up to 7 Days
  Frequency of presence of facial amimia versus non-amimia expressions between the groups.
Dynamic activity versus static position | Changes from Baseline up to 7 Days
  Percentage of time spent moving versus static position

CONTACTS AND LOCATIONS:
Overall Officials: Azra Bihorac, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No